CLINICAL TRIAL: NCT05217979
Title: Pulsed Radiofrequency Therapy for Hand OsteoArthritis Pain
Acronym: PROAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Margreet Kloppenburg, MD PhD, Professor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P21.101
Record Dates: First submitted 2021-12-17; First posted 2022-02-01 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Hand Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous pulsed radiofrequency (Active Comparator): After signing informed consent, patients assigned to the intervention group by randomization will receive a single treatment with transcutaneous pulsed radiofrequency.
  Interventions: Device: Transcutaneous pulsed radiofrequency
- Sham (Sham Comparator): After signing informed consent, patients assigned to the sham group by randomization will receive a single treatment with sham, which is indistinguishable from the active treatment. This is achieved by putting the device in demo mode, which gives all the same audiovisual signals as the active mode, but no treatment. Given that the treatment is not felt by patients, this ensures blinding.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Transcutaneous pulsed radiofrequency — single treatment with transcutaneous pulsed radiofrequency, for a duration of 15 minutes, at a strength of 800 mA.
  Arms: Transcutaneous pulsed radiofrequency
Device: Sham — Sham treatment by turning on the device in demo mode. No treatment delivered, but indistinguishable by sound or visual signals or sensations felt by the study participant
  Arms: Sham

SUMMARY:
Different types of pain may be present in patients with hand osteoarthritis, including nociceptive pain and non-nociceptive pain. This makes adequate pain treatment difficult, and thus new treatment options are needed. To this end, this trial will evaluate the effect of transcutaneous pulsed radiofrequency for the treatment of hand osteoarthritis pain.

DETAILED DESCRIPTION:
In this randomized clinical trial, patients with hand osteoarthritis, recruited from the Leiden University Medical Center Rheumatology outpatient clinic, aged 18-80 and fulfilling hand pain criteria will be randomized to undergo trancutaneous pulsed radiofrequency therapy of the hand or a sham. The effect will be measured in change in 10 point numeric rating scale for pain in the hand over 6 weeks. This RCT will have little burdens and risk for the subjects. The proposed intervention, tPRF, is well tolerated, with no known serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Hand osteoarthritis according to the ACR criteria
* Hand pain of at least 30mm on a 100mm VAS
* Chronic hand pain

Exclusion Criteria:

* Known inflammatory rheumatic diseases
* Psoriasis
* Seropositivity for rheumatoid factor of anti-CCP antibodies
* No understanding of the Dutch language
* Fibromyalgia (Following the ACR 2011 classification criteria)
* Neurological disorders interfering with pain perception and measurements
* Carpal tunnel syndrome interfering with pain perception and measurements
* History of chemo- and/or radiotherapy
* Spinal surgery or spinal trauma with lasting complaints interfering with pain perception and measurements
* Cognitive impairment or psychiatric conditions interfering with pain perception and measurements
* Pregnancy or breast-feeding
* Eye surgery for glaucoma or keratoconus or other surgery of the cornea in the three preceding months
* Presence of an implantable cardioverter-defibrillator (ICD), neurostimulator or pacemaker
* Metal implants in the hand, arm, shoulder or neck of the side that is to be treated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Hand pain at 6 weeks after trancutaneous pulsed radiofrequency or sham | 6 weeks
  Hand pain measured in a 0-10 numeric rating scale after trancutaneous pulsed radiofrequency or sham

SECONDARY OUTCOMES:
Hand pain at 12 weeks after trancutaneous pulsed radiofrequency or sham | 12 weeks
  Hand pain measured in a 0-10 numeric rating scale after trancutaneous pulsed radiofrequency or sham
Efficacy of transcutaneous pulsed radiofrequency on hand function | 6 weeks, 12 weeks
  Efficacy of trancutaneous pulsed radiofrequency on hand function (Australian/Canadian Hand Osteoarthritis Index [AUSCAN] function subscale, range 0-36, with higher scores indicating lower function)
Efficacy of transcutaneous pulsed radiofrequency on hand stiffness | 6 weeks, 12 weeks
  Efficacy of trancutaneous pulsed radiofrequency on hand stiffness (Australian/Canadian Hand Osteoarthritis Index [AUSCAN] stiffness subscale, range 0-4, with higher scores indicating more stiffness)
Efficacy of transcutaneous pulsed radiofrequency on the number of tender joints | 6 weeks, 12 weeks
  Efficacy of trancutaneous pulsed radiofrequency on the number of tender joints (Tender joint count)
Efficacy of trancutaneous pulsed radiofrequency on anxiety | 6 weeks, 12 weeks
  Efficacy of trancutaneous pulsed radiofrequency on anxiety measured with the Hospital Anxiety and Depression Scale, anxiety subscale, range 0-21, with higher scores indicating higher likeliness of anxiety, in patients with hand osteoarthritis
Efficacy of trancutaneous pulsed radiofrequency on depression | 6 weeks, 12 weeks
  Efficacy of trancutaneous pulsed radiofrequency on depression measured with the Hospital Anxiety and Depression Scale, depression subscale, range 0-21, with higher scores indicating higher likeliness of depression, in patients with hand osteoarthritis
Global perceived effect of recovery due to trancutaneous pulsed radiofrequency | 6 weeks, 12 weeks
  Global perceived effect of recovery due to trancutaneous pulsed radiofrequency, range 0-7, with lower scores indicating better outcomes, reported by patients with hand osteoarthritis
Global perceived effect of satisfaction with trancutaneous pulsed radiofrequency | 6 weeks, 12 weeks
  Global perceived effect of satisfaction with trancutaneous pulsed radiofrequency, range 0-7, with lower scores indicating better outcomes, reported by patients with hand osteoarthritis
Effect of transcutaneous pulsed radiofrequency therapy on health related quality of life | 6 weeks, 12 weeks
  Effect of transcutaneous pulsed radiofrequency therapy on health related quality of life measured with Short Form-36. Scores are standardized with a mean of 50 and sd of 10, with higher scores indicating better outcomes
Effect of transcutaneous pulsed radiofrequency therapy on temporal summation assessed using a 256 mN PinPrick | 6 weeks
  Effect of transcutaneous pulsed radiofrequency therapy on abnormalities measured with temporal summation, scored as present or absent. Patients will receive a single stimulation with the pinprick, scored 0-10 on NRS pain, followed by 10 stimuli with the pinprick, of which the last stimulus is scores 0-10 on NRS pain. This is repeated 5 times. The single stimuli are averaged, as are the 10th stimuli, and the ratio between these averages is calculated. A ratio >2 is indicative of temporal summation.
Effect of transcutaneous pulsed radiofrequency therapy on numbness of the hand. | 6 weeks
  Effect of transcutaneous pulsed radiofrequency therapy on numbness scored as present or absent, based on 5 stimuli with the PinPrick. Any stimulus rated as numb is regarded abnormal.
Effect of transcutaneous pulsed radiofrequency therapy on allodynia | 6 weeks
  Effect of transcutaneous pulsed radiofrequency therapy on allodynia, scored as present or absent. Scoring based on stimuli with a standardized brush, which is used to apply 5 stimuli to the back of the hand. Any of the stimuli evoking pain (score of >0 on a 0-10 NRS) is regarded as abnormal.
Effect of transcutaneous pulsed radiofrequency therapy on PainDETECT scores | 6 weeks, 12 weeks
  Effect of transcutaneous pulsed radiofrequency therapy on PainDETECT scores (range -1 to 38, with scores <13 indicating presence of neuropathic pain is unlikely, scores 13-18 indicating presence of neuropathic pain is undetermined and scores >18 indicating neuropathic pain presence is likely).
Effect of transcutaneous pulsed radiofrequency therapy on Michigan Hand Outcome Questionnaire | 6 weeks, 12 weeks
  Effect of transcutaneous pulsed radiofrequency therapy on MHOQ scores, ranged 0-100 per domain, with higher scores indicating better oucomes.
Effect of transcutaneous pulsed radiofrequency therapy on AUSCAN pain scores | 6 weeks, 12 weeks
  Effect of transcutaneous pulsed radiofrequency therapy on AUSCAN pain scores (Australian/Canadian Hand Osteoarthritis Index [AUSCAN] pain subscale, range 0-20, with higher scores indicating more pain)
Effect of transcutaneous pulsed radiofrequency therapy on central sensitization index scores | 6 weeks, 12 weeks
  Effect of transcutaneous pulsed radiofrequency therapy on central sensitization index scores, range 0-100, with higher scores indicating more signs of central sensitization.

OTHER OUTCOMES:
Effect of local inflammation at baseline on the efficacy of tPRF | 6 weeks, 12 weeks
  Effect of local inflammation at baseline as measured by ultrasonography based on power doppler signal, effusion and gray scale synovitis, on the efficacy of tPRF in reducing pain in hand osteoarthritis.
Effect of different QST profiles on tPRF efficacy | 6 weeks, 12 weeks
  Effect of different profiles based on quantitative sensory testing on tPRF efficacy in treating pain in hand osteoarthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Margreet Kloppenburg, Prof. Dr., Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No